CLINICAL TRIAL: NCT01196104
Title: A Phase 3b, Multicenter, Open-label, Randomized, Forced-titration Clinical Trial Evaluating the Efficacy and Safety of Technosphere® Insulin Inhalation Powder, Using the Gen2 Inhaler, in Combination With Insulin Glargine Versus Insulin Aspart in Combination With Insulin Glargine in Subjects With Type 2 Diabetes Mellitus Over a 16-week Treatment Period
Brief Title: Clinical Trial Evaluating the Efficacy and Safety of Technosphere® Inhalation Insulin (TI) Inhalation Powder Using the Gen2 Inhaler
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For Business Reasons
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-162
Record Dates: First submitted 2010-08-30; First posted 2010-09-08 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technosphere® Insulin Inhalation Powder (TI) (Experimental): Insulin Glargine and Technosphere® Insulin Inhalation Powder
  Interventions: Drug: Technosphere® Insulin Inhalation Powder; Drug: Insulin Glargine
- Comparator (Active Comparator): Insulin Glargine and Insulin Aspart
  Interventions: Drug: Insulin Aspart; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder
  Arms: Technosphere® Insulin Inhalation Powder (TI)
Drug: Insulin Aspart — Usual Care
  Arms: Comparator
Drug: Insulin Glargine

SUMMARY:
This is an open-label, randomized, forced-titration clinical trial evaluating the efficacy and safety of Technosphere Insulin (TI) Inhalation Powder in combination with insulin glargine versus insulin aspart in combination with insulin glargine in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Phase 3 clinical trial is designed to examine the efficacy and safety of inhaled prandial TI Inhalation Powder in combination with basal insulin verses insulin aspart in combination with basal insulin in subjects with type 2 diabetes who are suboptimally controlled with their current insulin regimens.This trial will employ a variety of methods to intensively manage these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 and ≤ 80 years of age
* Clinical diagnosis of type 2 diabetes mellitus for more than 12 months
* Body mass index (BMI) ≤ 45 kg/m2
* Glycated Hemoglobin (HbA1c) > 6.5% and ≤ 10.0%
* Treatment with 1 to 3 Oral Antidiabetic Drugs (OADs) and basal insulin for a minimum of 3 months before screening. Doses of OADs must have been stable for 3 months before study entry
* Nonsmokers (includes cigarettes, cigars, pipes, and chewing tobacco) for the preceding ≥ 6 months
* Office spirometry at the investigator site

  * Forced expiratory volume in 1 second (FEV1) ≥ 65% Third National Health and Nutrition Examination Survey (NHANES III) predicted
  * Forced vital capacity (FVC) ≥ 65% NHANES III predicted
  * Forced expiratory volume in 1 second as a percentage of forced vital capacity (FEV1/FVC) ≥ lower limit of normal (LLN)

Exclusion criteria:

* Current or prior treatment with prandial or PreMix (70/30) insulin
* History of insulin pump use within 6 weeks of Visit 1
* Treatment with Glucagon-like Peptide (GLP-1) analog drugs within the preceding 12 weeks of Visit 1
* History of chronic obstructive pulmonary disease (COPD), asthma, or any other clinically important pulmonary disease (eg, pulmonary fibrosis)
* Any clinically significant radiological findings on screening chest x-ray
* Use of medications for asthma, COPD, or any other chronic respiratory conditions
* Evidence of serious complications of diabetes (eg, symptomatic autonomic neuropathy)
* Significant cardiovascular dysfunction or history within 3 months of Visit 1 (eg, congestive heart failure [New York Heart Association {NYHA} Class III or IV])
* Serious arrhythmia, myocardial infarction, cardiac surgery, recurrent syncope, transient ischemic attacks, or any cerebrovascular accident
* History of pulmonary embolism or deep venous thrombosis in the 12 months before Screening (Visit 1)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Valley Research, Fresno, California
  - Health Care Partners Medical Group, Long Beach, California
  - Diabetes Research Center, Tustin, California
  - Diablo Clinical Research, Walnut Creek, California
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - John H Stoger Jr Hospital of Cook County, Chicago, Illinois
  - LaPorte County Institute for Clinical Research Inc., Michigan City, Indiana
  - Radiant Research Inc (Minneapolis), Edina, Minnesota
  - Amin Radparvar's Private Practice, City of Saint Peters, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - University of New Mexico HCS, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Endocrine Research Physicians East PA, Greenville, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - Legacy Clinical Research, Portland, Oregon
  - OHSU Diabetes Center Research Oregon Health & Science University, Portland, Oregon
  - The Endocrine Clinic, Memphis, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Exodus Healthcare Network, Magna, Utah
  - Diabetes Research Center -Fletcher Allen Health Care, South Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The FIrst Patient First Visit (FPFV) was September 21, 2010, and Last Patient Last Visit (LPLV) was August 25, 2011. Trial conducted in US. The study was terminated before completion of full enrollment for business reasons. Subjects already enrolled were allowed to complete the study to assess the safety of the titration algorithms.
Pre-assignment Details: After a 1 week to 5 week run-in period, subjects were randomized to receive either TI Inhalation Powder in combination with insulin glargine, or insulin aspart in combination with insulin glargine.
  105 Screened/46 Eligible. 39 subjects were randomized; 59 screen failures and 7 were screened but not randomized.
Groups:
- Technosphere Insulin + Insulin Glargine: Technosphere Insulin Inhalation Powder (administered prior to each meal) in combination with insulin glargine (once or twice daily); doses individualized for each patient
- Insulin Aspart + Insulin Glargine: Insulin Aspart (prior to each meal) and Insulin Glargine (once or twice daily) ; doses individualized for each patient
Period: Overall Study
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Started | 19 | 20
Completed | 15 | 15
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Various | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Full Range); unit: years] | 60.6 (7.95) [47 to 72] | 58.1 (10.67) [42 to 78] | 59.4 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37
Duration of Diabetes [Mean (Full Range); unit: years] | 14.6 (7.95) [3.7 to 35.9] | 15.6 (10.67) [2.5 to 43.1] | 15.1 [2.5 to 43.1]
Body Weight [Mean (Full Range); unit: kg] — Body Weight (kg) at Randomization
  kg | 100.9 (21.84) [54.1 to 141.9] | 100.8 (20.30) [66.4 to 138.6] | 100.9 [54.1 to 141.9]
Body Mass Index [Mean (Full Range); unit: kg/m2] — Body Mass Index (kg/m2) at Randomization
  kg/m2 | 33.2 (5.78) [19.3 to 42.9] | 33.3 (5.51) [24.3 to 44.1] | 33.2 [19.3 to 44.1]
HbA1c [Mean (Full Range); unit: %] — HbA1c (%) at randomization (NOTE: Aspart group only had 17 with HbA1c measurements at baseline)
  % | 7.76 (1.097) [6.3 to 10.2] | 7.94 (1.098) [6.7 to 10.3] | 7.85 [6.3 to 10.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (%) From Baseline to Week 16
Description: Change from Baseline in glycated hemoglobin at Week 16
Time Frame: Baseline to Week 16
Population: Safety Population, participants with data available at Baseline and Week 16
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of total hemoglobin
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 16 | 14
Percentage of total hemoglobin | -1.2179 (0.1468) | -1.2652 (0.1571)
Statistical Analysis 1: Comparison: Insulin Aspart + Insulin Glargine; ANCOVA model with terms of treatment as a fixed effect and baseline HbA1c as covariate; Test type: Non-Inferiority or Equivalence — Study terminated early due to business reasons, results are not properly powered; p = 0.8283, ANCOVA; Mean Difference (Final Values) = -0.0473, 95% CI 2-sided [-0.4901 to 0.3956], Standard Error of Mean 0.2158

2. Secondary Outcome: To Evaluate the Effect of Each Treatment on HbA1c
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Comparison of Fasting Plasma Glucose (FPG) Levels at Randomization and Throughout the Study
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Comparison of Post-prandial Glucose (PPG) Levels at Randomization and Throughout the Study
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Glycomark and Fructosamine Levels Measured Throughout the Study
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Seven-point Glucose at Randomization and Throughout the Study
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Glycemic Excursions and Variability as Assessed Through Continuous Glucose Monitoring (CGM)
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Body Weight at 16 Weeks
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Treatment Satisfaction as Assessed by Subject Treatment and Health Outcomes Questionnaires
Description: Not analyzed due to early termination of the trial.
Time Frame: Change from baseline to 16 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Total Number of Cough Episodes
Description: Total number of times patients coughed once, intermittently or continuously (inclusive)
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Cough episodes
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Cough episodes | 5 | 0

11. Secondary Outcome: Severe Hypoglycemic Event Rate
Description: Severe hypoglycemic event rate, ie, total number of events divided by subject-months of observation
  Severe hypoglycemia is defined as a subject who requires the assistance of another individual (not merely requested) and either:
  * SMBG levels ≤ 36 mg/dL OR
  * There is a prompt response to the administration of carbohydrate, glucagon, or other resuscitative measures
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Events / subject-month
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Events / subject-month | 0.01 | 0.34

12. Secondary Outcome: Mild or Moderate Hypoglycemic Event Rate
Description: Mild or moderate hypoglycemic event rate, ie, total number of events divided by subject-months of observation
  Nonsevere hypoglycemia is defined as a subject:
  * SMBG levels < 70 mg/dL AND/OR
  * Symptoms that are relieved by the self-administration of carbohydrates
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Events / subject-month
Groups:
- Technosphere® Insulin Inhalation Powder (TI): Insulin Glargine and Technosphere® Insulin Inhalation Powder
  Technosphere® Insulin Inhalation Powder
  Insulin Glargine
- Comparator: Insulin Glargine and Insulin Aspart
  Insulin Aspart: Usual Care
  Insulin Glargine
Arm/Group | Technosphere® Insulin Inhalation Powder (TI) | Comparator
Number analyzed (Participants) | 19 | 18
Events / subject-month | 4.47 | 4.41

13. Secondary Outcome: Number of Subjects Reporting Cough Episodes
Description: Number of Subjects Reporting Cough Episodes
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Number of participants
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Number of participants | 4 | 0

14. Secondary Outcome: Number of Subjects Reporting Intermittent Coughing Episodes
Description: Number of subjects reporting Intermittent Coughing Episodes
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Number of participants
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Number of participants | 4 | 0

15. Secondary Outcome: Number of Single Coughing Episodes
Description: Total number of times patients coughed only once
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Cough episodes
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Cough episodes | 1 | 0

16. Secondary Outcome: Number of Cough Episodes Occuring Within 10 Minutes of Drug Inhalation
Time Frame: Baseline to Week 16
Population: Safety Population
Measure: Number; unit: Cough episodes
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
Cough episodes | 5 | 0

17. Secondary Outcome: Baseline Forced Expiratory Volume in 1 Second (FEV1)
Description: Baseline FEV1
Time Frame: Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
L | 2.97 (0.63) | 2.83 (0.75)

18. Secondary Outcome: Week 16 Forced Expiratory Volume in 1 Second
Description: Week 16 FEV1
Time Frame: Week 16
Population: Safety Population, with data available at Week 16
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 14 | 15
L | 2.91 (0.57) | 2.66 (0.70)

19. Secondary Outcome: Week 16 Change From Baseline in Forced Expiratory Volume in 1 Second
Description: Week 16 Change from Baseline in FEV1
Time Frame: Baseline to Week 16
Population: Safety Population, with data available at Week 16
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 14 | 15
L | -0.14 (0.32) | -0.07 (0.27)

20. Secondary Outcome: Week 20 (Follow-up) Forced Expiratory Volume in 1 Second
Description: Week 20 (Follow-up) FEV1, 4 weeks after discontinuation of study treatment
Time Frame: Week 20 (Follow-up)
Population: Safety Population, with data available at Week 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 13 | 14
L | 3.07 (0.55) | 2.86 (0.70)

21. Secondary Outcome: Week 20 (Follow-up) Change From Baseline in Forced Expiratory Volume in 1 Second
Description: Week 20 (Follow-up, 4 weeks after discontinuation of study treatment) Change from Baseline in FEV1
Time Frame: Baseline to Week 20
Population: Safety Population, with data available at Week 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 13 | 14
L | -0.07 (0.29) | -0.05 (0.28)

22. Secondary Outcome: Baseline Forced Vital Capacity (FVC)
Description: Baseline FVC
Time Frame: Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 19 | 18
L | 3.63 (0.78) | 3.48 (1.02)

23. Secondary Outcome: Week 16 Forced Vital Capacity
Description: Week 16 FVC
Time Frame: Week 16
Population: Safety Population, with data available at Week 16
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 14 | 15
L | 3.61 (0.72) | 3.33 (0.98)

24. Secondary Outcome: Week 16 Change From Baseline Forced Vital Capacity
Description: Week 16 Change from Baseline FVC
Time Frame: Baseline to Week 16
Population: Safety Population, with data available at Week 16
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 14 | 15
L | -0.13 (0.34) | -0.07 (0.36)

25. Secondary Outcome: Week 20 (Follow-up) Forced Vital Capacity
Description: Week 20 (Follow-up, 4 weeks after discontinuation of study treatment) FVC
Time Frame: Week 20
Population: Safety Population, with data available at Week 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 13 | 14
L | 3.77 (0.73) | 3.57 (0.96)

26. Secondary Outcome: Week 20 (Follow-up) Change From Baseline in Forced Vital Capacity
Description: Week 20 (Follow-up, 4 weeks after discontinuation of study treatment) Change from Baseline in FVC
Time Frame: Baseline to Week 20
Population: Safety Population, with data available at Week 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Technosphere Insulin + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 13 | 14
L | -0.05 (0.35) | -0.06 (0.38)

ADVERSE EVENTS:
Time Frame: From first dose to 30d post last dose
Arm/Group | Technosphere® Insulin Inhalation Powder (TI) | Comparator
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18
Other Adverse Events (participants affected / at risk) | 13/19 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere® Insulin Inhalation Powder (TI) (N=19) | Comparator (N=18)
Angina unstable (Cardiac disorders) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Technosphere® Insulin Inhalation Powder (TI) (N=19) | Comparator (N=18)
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Mydriasis (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1
Ear Infection (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Blood Testosterone Decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cataract Operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
- Early termination of trial leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.